CLINICAL TRIAL: NCT00496717
Title: Measurement of an Abdominal Aorta Calcium Scoring and Its Correlation With Cardiovascular Risk Factors
Brief Title: Aorta Calcium Scoring
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Christine GEILLER, Directeur de la DRCI, University Hospital, Strasbourg, France
Other Study IDs: 3914
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-05

CONDITIONS: Cardiovascular Diseases
Keywords: Calcium scoring/aorta/ cardiovascular risk factor/scann; Patients with at least one cardiovascular risk factor
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: There is only one arm and all patients will have their aortic calcium scoring by CT scan.
  Interventions: Device: Helicoidal fast scann

INTERVENTIONS:
Device: Helicoidal fast scann — Each patient will have an computed aortic tomodensitometric scan without contrast injection. This procedure lasts few minutes and irradiation is low. The aortic calcium scoring is calculated using a specific program included in the scan machine

SUMMARY:
Calcium scoring of the coronary arteries is use as a predictor of coronary stenosis. The aim of this study is to measure the calcium scoring of the abdominal aorta using an helicoidal fast scan and to correlate this measurement with classical cardiovascular risk factors and newer parameters reflecting vascular rigidity, like pulse velocity measurement.

ELIGIBILITY:
Inclusion criteria :

* Patients with at least one cardiovascular risk factor
* Ambulatory or hospitalized patients

Exclusion criteria :

* Significant cardiovascular complications

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with at least one cardiovascular risk factor in primary prevention. Mainly out patients followed in our cardiology clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique STEPHAN, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (2):
- France (2):
  - Service d'Hypertension, Maladies Vasculaires et Pharmacologie Clinique, Nouvel Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Service de Radiologie, Hôpital Civil, Strasbourg